CLINICAL TRIAL: NCT05541380
Title: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients (TOPICS-THYROID)
Status: Active, not recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T2322
Record Dates: First submitted 2022-09-04; First posted 2022-09-15 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Thyroid Cancer
Keywords: advanced thyroid cancers; Registry Study
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. One H&E staining slide, and 10-18 tissue slides (5 um thickness) for cancer panel.
  2. Details of Tests/Collaborative Test Unit:
     Testing will take place in a certified precision medicine laboratory.
  3. Non-tumor Sample (Blood): Eight (8) ml of blood in EDTA tube will be collected from the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort A: patients who were pathologically (histologically) diagnosed as papillary carcinoma (PTC). They are in advanced stage and need systemic therapies. These patients may be unresectable, recurrent, persistent, or metastatic disease with RAI refractory or ineligible and need systemic therapies.
  Interventions: Other: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients
- Cohort B: patients who were pathologically diagnosed as DTC other than PTC, which includes follicular carcinoma, Hurthle cell carcinoma, and poorly differentiated carcinoma. The patients are in advanced stage and need systemic therapies. These patients may be unresectable, recurrent, persistent, or metastatic disease with RAI refractory or ineligible and need systemic therapies.
  Interventions: Other: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients
- Cohort C: patients who were pathologically diagnosed as medullary thyroid cancer (MTC) with persistent disease.
  Interventions: Other: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients
- Cohort D: patients who were pathologically diagnosed as anaplastic thyroid cancer (ATC).
  Interventions: Other: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients
- Cohort E: the patients who had performed large scale NGS oncopanel test previously and fulfil with the criteria in cohort A, B, C, or D.
  The patients must meet all the inclusion criteria and none of the exclusion criteria in each cohort.
  Interventions: Other: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients

INTERVENTIONS:
Other: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients — A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registry Study for Advanced Thyroid Cancer Patients

SUMMARY:
Because one cancer type may harbor various genetic aberrations, it is not enough to check only one or a few genes for a patient to choose the adequate treatment. Because the advance in multiplex genomic testing, several NGS-based cancer-associated genetic panel tests (oncopanel) have been developed and used to identify the genetic alterations, particularly the actionable genes, in each patient. Large scale checks of oncopanel have been executed in US. The study showed the genetic alterations in various cancer types and 11% of the patients had further molecular targeted therapy based on the result of the oncopanel test. Similar program was also conducted in Japan. Moreover, the oncopanel tests have been implicated in their clinical practice and the cost was reimbursed by the government of Japan and Korea recently. Precision medicine and such personalized treatment is the trend of cancer treatment. The trend of such treatment patterns is also observed in Taiwan. The genetic background for cancer treatment may also be different among different areas and races. There is short of genetic alteration data in Taiwanese cancer patients. To understand the landscape of genetic aberrations of cancer in Taiwan, large scale survey of the cancer patients is indicated. investigators propose to evaluate the landscape of genetic aberrations in cancer patients via oncopaenl test and collect the clinical data of the patients. The result of the oncopanel test will be provided to patients and their attending physicians as reference for their further treatment. In addition, investigators want to correlate the clinical outcome with the genetic aberrations of the cancer patients in Taiwan. Thyroid cancers are divided into differentiated thyroid cancer (DTC), medullary and anaplastic carcinoma. The majority of the patients are DTC. Different from other cancer type, radioactive iodine (RAI) therapy is usually the main treatment for advanced DTC. Multitargeted kinase inhibitors are indicated for advanced DTC refractory to RAI therapy and advanced medullary thyroid cancer. For anaplastic thyroid cancer, the prognosis is poor in spite of chemotherapy or radiation therapy. BRAF or NTRK targeted therapies are suggested if the patients have these genetic aberrations. Thyroid cancer patients have various genetic aberrations, including BRAF, RAS, RET, NTRK and others. Various gene specific kinase inhibitors have been developed and demonstrated the efficacy for the treatment of advanced thyroid cancer in addition to current standard therapies. Thyroid cancer is a cancer type with high percentage of driver gene aberration, however the genetic landscape of thyroid cancer is not well understood in Taiwan. In the current study, investigators want to investigate the genetic aberrations of advanced thyroid cancers by performing the NGS oncopanel.

DETAILED DESCRIPTION:
Cancer is the most common cause of death in Taiwan since 1982. The incidence of cancer is increasing worldwide, including Taiwan. Cancers in early stage can usually be treated by surgery with a good prognosis. However, the prognosis for recurrent, locally advanced or metastatic cancers is poor with a shorter survival. Systemic treatments are usually indicated for these patients. Chemotherapy is the mainstay for advanced cancer patients. However, the advances in the understanding of cancer biology and identification of targeted therapeutics not only increase the treatment strategies of cancer but also improve the survival and quality of life of the cancer patients. There are more and more molecularly targeted therapy developed and approved for the treatment of advanced cancer patients currently, which makes the beginning of precision cancer medicine. There are more and more treatments can be used based on the genetic aberrations of the cancers. Because one cancer type may harbor various genetic aberrations, it is not enough to check only one or a few genes for a patient to choose the adequate treatment. Because the advance in multiplex genomic testing, several NGS-based cancer-associated genetic panel tests (oncopanel) have been developed and used to identify the genetic alterations, particularly the actionable genes, in each patient. Large scale checks of oncopanel have been executed in US. The study showed the genetic alterations in various cancer types and 11% of the patients had further molecular targeted therapy based on the result of the oncopanel test. Similar program was also conducted in Japan. Moreover, the oncopanel tests have been implicated in their clinical practice and the cost was reimbursed by the government of Japan and Korea recently. Precision medicine and such personalized treatment is the trend of cancer treatment. The trend of such treatment patterns is also observed in Taiwan. The genetic background for cancer treatment may also be different among different areas and races. There is short of genetic alteration data in Taiwanese cancer patients. To understand the landscape of genetic aberrations of cancer in Taiwan, large scale survey of the cancer patients is indicated. investigators propose to evaluate the landscape of genetic aberrations in cancer patients via oncopaenl test and collect the clinical data of the patients. The result of the oncopanel test will be provided to patients and their attending physicians as reference for their further treatment. In addition, investigators want to correlate the clinical outcome with the genetic aberrations of the cancer patients in Taiwan. Thyroid cancers are divided into differentiated thyroid cancer (DTC), medullary and anaplastic carcinoma. The majority of the patients are DTC. Different from other cancer type, radioactive iodine (RAI) therapy is usually the main treatment for advanced DTC. Multitargeted kinase inhibitors are indicated for advanced DTC refractory to RAI therapy and advanced medullary thyroid cancer. For anaplastic thyroid cancer, the prognosis is poor in spite of chemotherapy or radiation therapy. BRAF or NTRK targeted therapies are suggested if the patients have these genetic aberrations. Thyroid cancer patients have various genetic aberrations, including BRAF, RAS, RET, NTRK and others. Various gene specific kinase inhibitors have been developed and demonstrated the efficacy for the treatment of advanced thyroid cancer in addition to current standard therapies. Thyroid cancer is a cancer type with high percentage of driver gene aberration, however the genetic landscape of thyroid cancer is not well understood in Taiwan. In the current study, investigators want to investigate the genetic aberrations of advanced thyroid cancers by performing the NGS oncopanel. Then investigators can understand the genetic aberrations of these patients in Taiwan and help search potential treatment targets for these patients.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

1. Pathologically confirmed papillary thyroid carcinoma (PTC).
2. The patient is in advanced stage, which includes recurrent, metastatic, unresectable, or persistent disease.
3. The patients are RAI-refractory* or ineligible for RAI therapy**.

   *The definitions of RAI-refractory are one of the following criteria: no uptake of RAI in the tumor, uptake of RAI in some tumors but no uptake in other tumors, disease progression in spite of RAI uptake in the tumors, or accumulated RAI dose ≥ 600 mCi.

   **the definitions of ineligible for RAI therapy are one of the following criteria: patients are unable to have RAI therapy due to some reasons, such as not received total thyroidectomy, unable to receive total thyroidectomy, or unable to have self-care in the isolation room.
4. The patient needs systemic therapy.
5. There are archived tumor samples available and the date of archived tumor sampling must be not more than 5 years from screening date. If there is no archived tumor sample available or the tumor sampling date is more than 5 years from screening date, re-biopsy is needed. If the quality of tumor sample is not fit for NGS oncopanel test, re-biopsy is needed.
6. Age ≥ the legal age.
7. Life expectancy greater than 6 months.
8. Capable of understanding and complying with the protocol requirements and signed informed consent.

Cohort B:

1. Pathologically confirmed differentiated thyroid cancer (DTC) other than PTC, which includes follicular thyroid cancer (FTC), Hurthle cell carcinoma, and poorly-differentiated thyroid cancer.
2. The patient is in advanced stage, which includes recurrent, metastatic, unresectable, or persistent disease.
3. The patients are RAI-refractory* or ineligible for RAI therapy**.

   *The definitions of RAI-refractory are one of the following criteria: no uptake of RAI in the tumor, uptake of RAI in some tumors but no uptake in other tumors, disease progression in spite of RAI uptake in the tumors, or accumulated RAI dose ≥ 600 mCi.

   **the definitions of ineligible for RAI therapy are one of the following criteria: patients are unable to have RAI therapy due to some reasons, such as not received total thyroidectomy, unable to receive total thyroidectomy, or unable to have self-care in the isolation room.
4. The patient needs systemic therapy.
5. There are archived tumor samples available and the date of archived tumor sampling must be not more than 5 years from screening date. If there is no archived tumor sample available or the tumor sampling date is more than 5 years from screening date, re-biopsy is needed. If the quality of tumor sample is not fit for NGS oncopanel test, re-biopsy is needed.
6. Age ≥ the legal age.
7. Life expectancy greater than 6 months.
8. Capable of understanding and complying with the protocol requirements and signed informed consent.

Cohort C:

1. Pathologically confirmed medullary thyroid carcinoma (MTC).
2. The patient is in advanced stage, which includes recurrent, metastatic, unresectable, or persistent disease.
3. There are archived tumor samples available and the date of archived tumor sampling must be not more than 5 years from screening date. If there is no archived tumor sample available or the tumor sampling date is more than 5 years from screening date, re-biopsy is needed. If the quality of tumor sample is not fit for NGS oncopanel test, re-biopsy is needed.
4. Age ≥ the legal age.
5. Life expectancy greater than 6 months.
6. Capable of understanding and complying with the protocol requirements and signed informed consent.

Cohort D:

1. Pathologically confirmed anaplastic thyroid carcinoma (ATC).
2. There are archived tumor samples available and the date of archived tumor sampling must be not more than 5 years from screening date. If there is no archived tumor sample available or the tumor sampling date is more than 5 years from screening date, re-biopsy is needed. If the quality of tumor sample is not fit for NGS oncopanel test, re-biopsy is needed.
3. Age ≥ the legal age.
4. Capable of understanding and complying with the protocol requirements and signed informed consent.

Cohort E:

The patients who had performed large NGS oncopanel test (ACTOnco) previously meet all the inclusion criteria of cohort A, B, C or D except the criteria of archived tumor sample requirement. These patients do not need to take archived tumor sample for NGS oncopanel test but need to take archived tumor sample for TERT promoter mutation and peripheral blood sampling.

-

Exclusion Criteria:

Cohort A:

1. Inability and unwillingness to give informed consent.
2. The patients have no evidence of disease before systemic treatment.
3. The patients have stable residual disease or metastatic disease without progression and do not need systemic therapies.
4. The patients do not intend to have systemic therapies.
5. Patients do not agree to provide archived tumor samples and blood samples or they do not agree to do tumor biopsy when archived tumor samples are not available or inadequate for NGS oncopanel test.
6. The date of archived tumor sampling is more than 5 years from screening date.
7. Patients refuse for collection of clinical data and follow-up.
8. Mental status is not fit for further treatment or data collection.

Cohort B:

1. Inability and unwillingness to give informed consent.
2. The patients have no evidence of disease before systemic treatment.
3. The patients have stable residual disease or metastatic disease without progression and do not need systemic therapies.
4. The patients do not intend to have systemic therapies.
5. Patients do not agree to provide archived tumor samples and blood samples or they do not agree to do tumor biopsy when archived tumor samples are not available or inadequate for NGS oncopanel test.
6. The date of archived tumor sampling is more than 5 years from screening date.
7. Patients refuse for collection of clinical data and follow-up.
8. Mental status is not fit for further treatment or data collection.

Cohort C:

1. Inability and unwillingness to give informed consent.
2. The patients have no evidence of disease before systemic treatment.
3. Patients do not agree to provide archived tumor samples and blood samples or they do not agree to do tumor biopsy when archived tumor samples are not available or inadequate for NGS oncopanel test.
4. The date of archived tumor sampling is more than 5 years from screening date.
5. Patients refuse for collection of clinical data and follow-p.
6. Mental status is not fit for further treatment or data collection.

Cohort D:

1. Inability and unwillingness to give informed consent.
2. Patients do not agree to provide archived tumor samples and blood samples or they do not agree to do tumor biopsy when archived tumor samples are not available or inadequate for NGS oncopanel test.
3. The date of archived tumor sampling is more than 5 years from screening date.
4. Patients refuse for collection of clinical data and follow up.

Cohort E:

The patients do not meet all exclusion criteria of cohort A, B, C, or D except for providing archived tumor sample.

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to include 250 advanced thyroid cancer patients, including 150 papillary thyroid cancer cancers (cohort A), and 50 non-PTC DTC, including follicular thyroid cancers, Hurthle cell carcinoma and poorly-differentiated carcinoma (cohort B), 25 medullary thyroid cancer (cohort C), and 25 anaplastic thyroid cancer (cohort D) in this study. There is no case number limitation for cohort E. However, we estimate to enroll approximately 50 patients in cohort E. In cohort A, the enrolled number of men and women must be ≥ 50 for each group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the genetic profiles in advanced thyroid cancer patients in Taiwan. | 5 years
  ACTonco+ACTFusion

CONTACTS AND LOCATIONS:
Locations (9):
- Taiwan (9):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District